CLINICAL TRIAL: NCT06950827
Title: Textbook Outcomes of Right Hemihepatectomy in Patients With Hepatocellular Carcinoma: a Comparative Study of Laparoscopic and Open Surgery
Brief Title: Textbook Outcomes of Right Hemihepatectomy in Patients With Hepatocellular Carcinoma
Status: Recruiting | Type: Observational
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Jiwei Huang, Clinical Professor, West China Hospital
Other Study IDs: JHuang20232
Record Dates: First submitted 2025-04-22; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Hepatocellular Carcinoma; Hepatectomy; Laparoscopic Hepatectomy
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hepatocellular carcinoma patients who received laparoscopic right hemihepatectomy
  Interventions: Procedure: laparoscopic right hemihepatectomy
- Hepatocellular carcinoma patients who received open right hemihepatectomy

INTERVENTIONS:
Procedure: laparoscopic right hemihepatectomy — Laparoscopic surgery has many advantages, such as small surgical incision and fast postoperative recovery. In recent years, more and more centers have gradually transitioned to performing right hemihepatectomy through laparoscopy as much as possible.
  Groups: Hepatocellular carcinoma patients who received laparoscopic right hemihepatectomy

SUMMARY:
Although traditional open right hemihepatectomy is a mature technique, the incision is usually very large; Intraoperative bleeding may be excessive, and postoperative liver failure is also prone to occur. In recent years, compared with traditional open surgery, laparoscopic surgery has many advantages, such as smaller surgical incision and faster postoperative recovery. In recent years, more and more centers have gradually transitioned to performing right hemihepatectomy through laparoscopy as much as possible. However, due to the difficulty of the surgery, steep learning curve, and postoperative complications, its adoption is limited to high-capacity surgical centers. Despite significant progress in laparoscopic liver resection technology, its clinical efficacy remains controversial, especially in laparoscopic right hemihepatectomy. More research is needed to confirm the feasibility and safety of this surgery. At present, it is unclear whether there is a difference in textbook outcomes (TO) between HCC patients undergoing open and laparoscopic right hemihepatectomy, and the association between TO and patient survival prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old;
2. The lesion is limited to the right half of the liver and diagnosed as hepatocellular carcinoma based on paraffin pathology and immunohistochemistry results;
3. The type of surgery is elective surgery;
4. The patient's preoperative liver function was Child Pugh A or B grade, and the preoperative ASA (American Society of Anesthesiologists) rating was I, II, or III.

Exclusion Criteria:

1. Pathological confirmed cholangiocarcinoma, mixed cell carcinoma, or extrahepatic metastatic malignant tumors;
2. Previous history of upper abdominal surgery;
3. Simultaneously undergoing adjacent abdominal organ resection, major vessel and biliary reconstruction surgery, except for the gallbladder;
4. Merge adjacent organ invasions except for the gallbladder, with main blood vessels, bile duct cancer emboli, or distant metastases;
5. Lost to follow-up or loss of primary clinical data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The data was collected from patients who underwent right hemihepatectomy and were diagnosed with HCC pathologically. The data was collected from the division of Liver Surgery of West China Hospital, SCU from January 2018 to January 2023.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-04-05 (Actual); Primary Completion 2025-05-10 (Estimated); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
Textbook outcome | From January 2018 to January 2023
  Textbook outcome (TO) was defined as the absence of intraoperative grade ≥ 2 incidents (defined according to the Oslo classification), postoperative bile leak of grade B or C (according to the severity grading of the International Study Group of Liver Surgery), postoperative liver failure grade B or C (according to the severity grading of the International Study Group of Liver Surgery), major postoperative complications within 90 days (Clavien-Dindo grade III or higher), readmission within 90 days after discharge due to surgery related major complications (Clavien-dindo Grade III or higher), in-hospital or 90-day mortality and the presence of R0 resection margin (i.e. 1mm or more tumor free margin).

SECONDARY OUTCOMES:
Overall survival | From January 2018 to January 2023
  Overall survival (OS) was defined as the interval from liver resection to death or the last follow-up.
Disease-free survival | From January 2018 to January 2023
  Disease-free survival (DFS) was defined as the time from liver resection to disease recurrence or death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No